CLINICAL TRIAL: NCT05036434
Title: A Prospective Phase II Trial of Pembrolizumab Plus Lenvatinib in Advanced Adrenal Cortical Carcinoma After Failure of Platinum- and Mitotane-Based Chemotherapy
Brief Title: Phase II Trial of Pembrolizumab Plus Lenvatinib in Advanced Adrenal Cortical Carcinoma
Acronym: ACCOMPLISH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: MSD Korea Ltd. (Industry)
Responsible Party: Principal Investigator, Tak Yun, Doctor of Medicine, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCT-STRC-02
Record Dates: First submitted 2021-08-26; First posted 2021-09-05 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Adrenocortical Carcinoma
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Pembrolizumab 200mg q 3wks IV / Lenvatinib 20mg daily once PO q 3wks
  Interventions: Drug: Pembrolizumab / Lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab / Lenvatinib — Pembrolizumab Plus Lenvatinib administration.
  Other Names: Keytruda / Lenvima

SUMMARY:
* Clinical Indication : Advanced adrenal cortical carcinoma after platinum-based chemotherapy
* Trial Type : Single arm, prospective trial
* Route of administration : Intravenous (pembrolizumab) and peroral (lenvatinib)
* Treatment Groups : Single arm
* Number of trial participants : 30

DETAILED DESCRIPTION:
1. Timing of Dose Administration for Pembrolizumab Trial interventions should be administered on Day 1 of each cycle after all procedures/assessments have been completed as detailed on the Schedule. Trial interventions may be administered up to 3 days before or after the scheduled Day 1 of each cycle due to administrative reasons.

   All trial interventions will be administered on an outpatient basis. Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks. Sites should make every effort to target infusion timing to be as close to 30 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -5 minutes and +10 minutes is permitted (i.e., infusion time is 30 minutes: -5 min/+10 min).
2. Lenvatinib administration Lenvatinib will be administered with water orally once a day (with or without food) in 21-day cycles at approximately the same time each day. Treatment cycles will be counted continuously regardless of dose interruptions. On Day 1 (D1) of each cycle, it will be administered approximately 1 hour after completion of pembrolizumab administration.
3. Treatment Period The Treatment Phase will begin with the administration of the first dose of study treatment to the first subject in Cycle 1 and continues in 21-day (3-week) cycles. Subjects will continue to receive study treatment until confirmed PD by IIR, development of unacceptable toxicity, subject request, withdrawal of consent, completion of 35 treatments (approximately 2 years) with pembrolizumab, or study termination by the sponsor. Those subjects that discontinue study treatment transition to the Off-Tx Visit of the Follow-up Period.
4. Safety Follow-Up Visit The mandatory Safety Follow-Up Visit should be conducted approximately 30 days after the last dose of study intervention or before the initiation of a new anti-cancer treatment, whichever comes first.
5. Efficacy Follow-up Visits Participants who complete the protocol-required cycles of study intervention of who discontinue study intervention for a reason other than disease progression will begin the Efficacy Follow-Up Phase and should be assessed every 6 weeks (42 ± 7 days) by radiologic imaging to monitor disease status. After 6 months, the imaging time point will occur every 9 weeks (± 7 days). Every effort should be made to collect information regarding disease status until the start of new anti-cancer therapy, disease progression, death, end of the study. Information regarding post-study anti-cancer treatment will be collected if new treatment is initiated. Participants who completed all efficacy assessments and/or will not have further efficacy assessments must enter the Survival Follow-up Phase.
6. Time Period and Frequency for Collecting AE, SAE, and Other Reportable Safety Event Information :

All AEs, SAEs, and other reportable safety events that occur after the consent form is signed but before intervention allocation must be reported by the investigator if the event cause the participant to be excluded from the study, or is the result of a protocol-specified intervention, including but not limited to washout or discontinuation of usual therapy, diet, or a procedure.

* All AEs from the time of intervention allocation through 30 days following cessation of study intervention must be reported by the investigator.
* All AEs meeting serious criteria, from the time of intervention allocation through 90 days following cessation of study intervention or 30 days following cessation of study intervention if the participant initiates new anticancer therapy, whichever is earlier, must be reported by the investigator.
* All pregnancies and exposure during breastfeeding, from the time of intervention allocation through 120 days following cessation of study intervention, or 30 days following cessation of study intervention if the participant initiates new anticancer therapy must be reported by the investigator.
* Additionally, any SAE brought to the attention of an investigator at any time outside of the time period specified above must be reported immediately to MSD if the event is considered drug-related.

Investigators are not obligated to actively seek AEs or SAEs or other reportable safety events in former study participants. However, if the investigator learns of any SAE, including a death, at any time after a participant has been discharged from the study, and he/she considers the event to be reasonably related to the study intervention or study participation, the investigator must promptly notify MSD.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 19 years of age on the day of signing informed consent with histologically confirmed diagnosis of adrenal cortical carcinoma will be enrolled in this study.
2. Patients with locally advanced, recurrent, or metastatic disease not amenable to surgery, radiotherapy, or combined modality therapy with curative intent.
3. Patients who have received prior systemic therapy including combined mitotane and cisplatin-based chemotherapy as a palliative aim systemic therapy in advanced setting, and have had disease progression within 6 months of the last dose of the most recent systemic therapy. Patients who discontinued prior therapy due to intolerable toxicities can be included.

   *However, patients who have not received prior mitotane therapy due to inability to import mitotane domestically who disease has progression may be exceptionally eligible for registration.
4. Patients should have measurable disease according to RECIST v1.1 meeting the following criteria:

   1. at least 1 lesion of ≥10 mm in the longest diameter for a non-lymph node or ≥15 mm in the short-axis diameter for a lymph node that is serially measurable according to RECIST using CT or MRI
   2. lesions that have had external beam radiotherapy or other loco-regoinal therapies such as radiofrequency ablastion must show subsequent evidence of substantial size increase to be deemed a target lesion.
5. Subject must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 1
6. Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP≤150/90 mmHg at screening and no change in hypertensive medications within 1 week prior to the cycle 1 day 1.
7. Adequate renal function defined as creatinine ≤1.5 times the upper limit of normal (×ULN) or calculated creatinine clearance ≥30 ml/min per the Cockcroft and Gault formula
8. Adequate bone marrow function:

   1. Absolute neutrophil count (ANC)≥1500/mm3 (≥1.5×103/μL)
   2. platelets≥100,000/ mm3 (≥100×109/L)
   3. hemoglobin≥9.0 g/dL
9. adequate blood coagulation function defined by international Normlized Ratio (INR)≤1.5 unless participant is receiving anticoagulation therapy
10. adequate liver function defined by:

    1. total bilirubin ≤1.5×ULN except for unconjugated hyperbilirubinemia of Gilbert's syndrome
    2. alkaline phosphatase (ALP), alanine aminotransferase (ALT), and asparate aminotransferase (AST)≤3×ULN (in the case of liver metastases ≤5×ULN), unless there are bone metastases. Subject with ALP values >3×ULN and known to have bone metastases can be included.
11. Life expectancy more than 3 months
12. Patients should agree to discontinue mitotane
13. Females of childbearing potential must agree to use a highly effective method of contraception for the entire study period and for 120 days after study discontinuation (see appendix 7)
14. Male participants who are partners of women of childbearing potential must use a condom plus spermicide and their female partners if of childbearing potential must use a highly effective method of contraception (see inclusion criterion #14 and appendix 7) beginning at least 1 mentrual cycle prior to starting study drugs, throughout the entire study period, and for 120 days after the last dose of study drug, unless the male subjects are totally sexually abstinent or have undergone a successful vasectomy with confirmed azoospermia or unless the female partners have been sterilized surgically or are otherwise proven sterile.
15. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated for biomarker analysis. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue. In the case of archival tissue cannot be provided, patients with inaccessible tumors for biopsy specimens or patients who refuse to be biopsied can be enrolled without a biopsy at the discretion of treating physician.
16. Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.
17. Participants who are HBsAg positive are eligible if they have received HBV anti-viral therapy for at least 4 weeks, and have undetectable HBV viral load.

Note: Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.

Participants with a history of HCV infection are eligible if HCV viral load is undetectable at screening Note: Participants must have completed curative anti-viral therapy at least 4 weeks prior to randomization.

Exclusion Criteria:

1. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
2. Has received prior therapy with any VEGFR TKI or monoclonal antibody targeting VEGF pathway.
3. Has received major surgery within 2 weeks of start of study intervention. Participants must have recovered from any toxicity and/or complications from major surgery prior to starting therapy.
4. Previous radiotherapy to the only measurable lesion: but previous radiotherapy will be permitted unless the lesion is the only measurable lesion.
5. Subjects having >1+ proteinuria on urinalysis will undergo 24-hour urine collection for quantitative assessment of proteinuria. Subjects with urine protein ≥1g/24-hour will be ineligible.
6. Gastrointestinal malabsorption, gastrointestinal obstruction, or any other condition that might affect the absorption of lenvatinib.
7. Significant cardiovascular impairment within 6 months of the first dose of study drug. History of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke, cardiac arrhythmia associated with significant cardiovascular impairment, or a left ventricular ejection fracture (LVEF) below the institutional normal range as determined by MUGA or echocardiogram.
8. Prolongation of QTc interval to >480 msec
9. Bleeding or thrombotic disorders or subjects at risk for severe hemorrhage. The degree of tumor invasion/infiltration of major blood vessels should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy.
10. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
11. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
12. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug. The use of physiologic doses of corticosteroids may be approved at the discretion of treating physician. In mitotane treated subject, adrenal insufficiency happens inevitably and required dose of corticosteroid is higher than usual due to altered metabolism of corticosteroid.48 Therefore, the decision on whether the dose of maintenance corticosteroid is acceptable for enrollment depends on investigator.
13. Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded. Clinically insignificant or curatively treated localized prostate cancer and curatively treated thyroid cancer of any stage can be included at the discretion of treating physician.
14. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
15. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
16. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis. Non-infectious pneumonitis include, but not limited to, idiopathic pulmonary fibrosis, organizing pneumonia, or drug-induced pneumonitis. History of radiation pneumonitis in the radiation field is permitted.
17. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
18. Has an active tuberculosis. However, inactive tuberculosis (previously treated or latent infection without evidence of active disease) is allowed.
19. Has a known history of Human Immunodeficiency Virus (HIV) infection.
20. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
21. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
22. All females with child-bearing capacity who has a positive urine pregnancy test within 72 hours prior to the first dose of study drug. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
23. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
24. Has had an allogenic tissue/solid organ transplant.
25. Serious nonhealing wound, ulcer, or bone fracture.
26. Has active infections that requires systemic therapy.
27. Has the side effect by previous treatment that has not recovered to baseline or below G1.
28. Has a known severe hypersensitivity reaction history of humanized monoclonal antibodies or VFGFR TKI including ingredients used in medication.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
To assess the antitumor activity of pembrolizumab plus lenvatinib in patients with advanced ACC. | Treatment-Related Adverse Events as Assessed by CTCAE v4.0, Imaging assessment by RECIST v1.1.
  Through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Tak Yun, Principal Investigator — National Cancer Center, Republic of Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea